CLINICAL TRIAL: NCT07037186
Title: Impact of Diabetes on Burst-Suppressions During Intraoperative EEG in Elderly Patients: Correlation With Postoperative Delirium
Brief Title: Burst Suppressions in Diabetic Elderly
Status: Active, not recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 30-2024
Record Dates: First submitted 2025-06-10; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Geriatric; General Anaesthesia; Electroencephalography; Oxymetry
Keywords: postoperative delirium; elderly; electroencephalography; burst suppression; diabetes mellitus; general anesthesia
MeSH Terms: conditions — Diabetes Mellitus; Emergence Delirium | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- DM-OAD: Diabetic patients who are under oral anridiabetic medcation and not used insulin regimens
  Interventions: Device: Electroencephalogram
- DM-Insulin: Diabetic patients under insulin regimen
  Interventions: Device: Electroencephalogram
- Non-DM: Patients without diabetes mellitus
  Interventions: Device: Electroencephalogram

INTERVENTIONS:
Device: Electroencephalogram — All patients will receive intraoperative electroencephalography monitorization during general anesthesia.

SUMMARY:
This observational study aims to learn about the effects of diabetes mellitus in intraoperative electroencephalography (EEG) of elderly patients receiving general anesthesia. The main question it seeks to answer is:

Is there a relation between preoperative diabetes, intraoperative electroencephalogram suppression ratio, and postoperative delirium?

Participants aged over 65, receiving general anesthesia as part of their anesthesia plan for surgery of any kind, will be monitored with EEG and cerebral oximetry intraoperatively to record burst suppressions and questioned for delirium for 48 hours postoperatively.

DETAILED DESCRIPTION:
3 different patient groups will be observed: those who are diagnosed with diabetes and use oral antidiabetics, those who receive insulin therapy with a diagnosis of diabetes, and patients whose preoperative fasting glucose values are confirmed to be normal without a diagnosis of diabetes.

Patients over 65 who are scheduled for any surgery requiring general anesthesia for at least 30 minutes will be evaluated to detect their basal cognition status with a mini-cognition test and a preoperative anesthesia examination. In addition to routine monitoring, this patient group will also be monitored with electroencephalogram and cerebral oximetry.

Anesthesia induction and maintenance for each patient are applied according to the values here. In the maintenance of anesthesia, sevoflurane will be regulated according to 0.7-1 MAC (adjusted for age), and remifentanil infusion will be regulated according to PSI. Postoperative analgesia will be achieved with tramadol 1 mg/kg and Parol 10 mg/kg (IV) with a target pain score below 4. Each patient will be evaluated with a NUDESC score as a delirium score in the postoperative PACU and during 48 hours in the ward. Values such as suppression time and ratio, the subject of study in EEG recordings during anesthesia, can only be seen by transferring them to the computer with a transfer cable, so the evaluations will be blind. All data transfers will be done after the 48th hour.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 65 undergoing ASA I-IV receiving general anaesthesia
* All elective surgery patients who are not laparoscopic and last longer than 30 minutes

Exclusion Criteria:

* 1) American Society of Anesthesiologists (ASA) grade V or VI
* Whether the surgery is cranial or laparoscopic
* Preoperative neuropsychiatric (dementia, epilepsy, etc.) disease or drug use
* Previous cranial surgery or known vertebrobasilar insufficiency, carotid stenosis
* Those with a pain score above 4 in the postoperative evaluation unit (PACU)
* Patients with a 15% decrease in cerebral oxygenation from onset in oximetry monitoring during follow-up
* Patients with bleeding greater than 20% of total body volume during follow-up
* Patients with a decrease of more than 20% from their baseline systolic value (based on follow-up in the service) during follow-up
* Those with hypercarbia or hypocarbia due to intraoperative ventilation insufficiency
* Patients whose PSI value is reduced to a depth of 25, which is sufficient for anaesthesia, with anaesthetic drugs administered during anaesthesia induction or maintenance
* Presence of preoperative cognitive dysfunction
* Patients requiring postoperative intubation and intensive care follow-up

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly patients receiving general anesthesia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
burst-suppression | Perioperative
  Burst suppression amount recorded during EEG monitorization under general anesthesia

SECONDARY OUTCOMES:
delirium | Perioperative
  postoperative delirium scanned with the nursing delirium screening scale (NUDESC)

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, MD, Study Chair — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Li A, Wang S, Wang T, Liu T, Wang Y, Fu J, Zhao G, Yang Q, Dong H. Differences in the EEG Power Spectrum and Cross-Frequency Coupling Patterns between Young and Elderly Patients during Sevoflurane Anesthesia. Brain Sci. 2023 Jul 31;13(8):1149. doi: 10.3390/brainsci13081149. PMID 37626505
- [Background] Shang Z, Jiang Y, Fang P, Zhu W, Guo J, Li L, Liang Y, Zhang S, Ma S, Mei B, Fan Y, Xie Z, Shen Q, Liu X. The Association of Preoperative Diabetes With Postoperative Delirium in Older Patients Undergoing Major Orthopedic Surgery: A Prospective Matched Cohort Study. Anesth Analg. 2024 May 1;138(5):1031-1042. doi: 10.1213/ANE.0000000000006893. Epub 2024 Feb 9. PMID 38335150